CLINICAL TRIAL: NCT04713644
Title: Study of the Association Between Burst Suppression During Anesthetic Induction With Propofol in Cardiac Surgery in Patients Over 65 Years of Age With Postoperative Delirium
Brief Title: Association Between Burst Suppression During Anesthetic Induction With Postoperative Delirium in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 200923005
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Delirium
Keywords: Burst Suppression; Postoperative Delirium; Electroencephalography; Propofol; Cardiac Surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C-reactive protein (CRP) serum level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Burst Suppression: Patients who present burst suppression after standardized propofol administration during anesthetic induction
  Interventions: Drug: Standardized Propofol Administration
- No Burst Suppression: Patients who did not present burst suppression after standardized propofol administration during anesthetic induction
  Interventions: Drug: Standardized Propofol Administration

INTERVENTIONS:
Drug: Standardized Propofol Administration — Intravenous bolus propofol administration of 0.5 mg/Kg dose, plus 0.5 mg/Kg extra if necessary

SUMMARY:
The population over 65 years of age will be increasingly exposed to surgical procedures that require general anesthesia. Postoperative delirium is one of the main causes of preventable postoperative morbidity in the elderly population and is a frequent event after cardiac surgery with extracorporeal circulation. The excess administration of anesthetics that potentiate the Gamma Aminobutyric A receptor, such as propofol, are related to an intraoperative electroencephalographic pattern called burst suppression that has been associated with postoperative delirium. It is unknown whether this pattern is secondary to a relative overdose of anesthetics or rather corresponds to a characteristic of a vulnerable brain that is suppressed at doses at which other patients are not. Our objective will be to determine whether burst suppression in people over 65 years of age during a standardized anesthetic induction with propofol for cardiac surgery with extracorporeal circulation is associated with postoperative delirium compared to older people who do not present it.

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders, including postoperative delirium (POD), are the leading cause of preventable postoperative morbidity in the elderly population. POD is an acute brain dysfunction characterized by changes in attention and cognition usually within of the first week after surgery and anesthesia. Its appearance triggers a series of events that often end in loss of independence, increased morbidity and mortality and increased health costs. It has been associated with the development of long-term cognitive impairment, including persistent dementia. Its nature is multifactorial and its pathophysiology is not yet fully elucidated.

Over administration of anesthetics that potentiate the Gamma Amino Butyric A (GABAA) receptor, such as barbiturates or propofol, is related to an intraoperative electroencephalographic (EEG) pattern called burst suppression that has been associated with POD. It is a common event after cardiac surgery with an incidence ranging from 15% to 50%. Given its adverse impact on functioning and quality of life, delirium has enormous social implications for the individual, family, community, and health care systems.

Burst suppression is a pattern observed in the EEG characterized by quasi-periodic alternations between isoelectricity (flat EEG) and brief bursts of electrical activity such as spikes, sharp waves, or slow waves. It reflects a brain state of relative cortical inactivity that is not observed during normal waking states or sleeping behaviors. This pattern can be observed associated with coma due to diffuse anoxic damage, induced hypothermia and Ohtahara syndrome epilepsy. In addition, the administration of high-dose anesthetics that potentiate the GABAA receptor produce burst suppression followed by isoelectricity. Burst suppression during maintenance of general anesthesia with anesthetics that enhance the GABAA receptor has previously been associated with POD. When propofol is administered as a bolus during anesthetic induction, older patients, can suffer burst suppression in seconds. However, it is unknown whether this pattern is secondary to a relative overdose of anesthetics or rather corresponds to a characteristic of the vulnerable brain that is suppressed at doses to which other patients do not present this pattern. At present, it is not known whether burst suppression is a modifiable risk factor for POD or an epiphenomenon or marker of other factors that cause POD. A randomized controlled clinical trial studied an EEG-guided anesthetic protocol that reduced the administration of anesthetic, diminished the incidence of burts suppression during the intraoperative period, but not the incidence of POD. Therefore, the association between bursts suppression induced by anesthetics and POD appears not to be causal.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years of age
* Undergoing elective cardiac surgery requiring extracorporeal circulation (coronary artery bypass, univalvular replacement, bivalvular and coronary artery bypass plus univalvular replacement)
* American Society of Anesthesiologists Physical Status II-III.

Exclusion Criteria:

* Body Mass Index > 35 and <18 Kg / m2
* Severe ventricular dysfunction (EF < 30% or severe dysfunction measured in ventriculography)
* Emergency surgery
* Chronic use of alcohol or drug abuse
* History of Stroke
* Neurological diseases
* Endocarditis
* Positive screening for preoperative delirium.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years of age undergoing cardiac surgery with cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Delirium | Up to 72 hours after surgery (3 postoperative days), CAM or CAM-ICU assessed twice daily (AM/PM)
  Positive Confusion Assessment Method (CAM), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), or structured chart review

SECONDARY OUTCOMES:
Burst suppression during anesthesia induction | 20 minutes after standardized propofol administration
  Burst suppression incidence after standardized propofol induction in patients ≥ 65 years scheduled for cardiac surgery with cardiopulmonary bypass
Burst suppression during cardiopulmonary bypass | Through Cardiopulmonary bypass time defined as time between connection to pump to disconnection, an average of 120 minutes
  Burst suppression incidence during cardiopulmonary bypass in patients ≥ 65 years scheduled for cardiac surgery with cardiopulmonary bypass
Preoperative Cognitive Status | Preoperative anesthetic evaluation
  Preoperative cognitive assessment using MiniCog, minimum value: 0 - maximum value:5 , higher scores meaning better outcomes. If MiniCog ≤ 2, MoCA (Montreal Cognitive Assessment) exam will be performed.
Preoperative Frailty | Preoperative anesthetic evaluation
  Preoperative frailty evaluation using Clinical Frailty Scale (CFS), minimum value: 1(Very Fit) - maximum value: 9 (Terminally Ill), higher scores meaning worse outcomes
Electroencephalogram (EEG) Alpha Power/Total Power | Stable anesthetic period before cardiopulmonary bypass and 20 minutes after propofol induction
  Electroencephalogram power between 8 to 12 Hz (Alpha) and 0.1 to 35 Hz (Total)
CRP (C Reactive Protein) | Blood sample collection during arterial line insertion, before anesthetic induction
  Serum C Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pedemonte, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
All data will be collected and saved in digital forms. Data may be shared with other researchers with previous authorization from the PI.

REFERENCES:
- [Background] Soreide K, Wijnhoven BP. Surgery for an ageing population. Br J Surg. 2016 Jan;103(2):e7-9. doi: 10.1002/bjs.10071. No abstract available. PMID 26771471
- [Background] Deiner S, Westlake B, Dutton RP. Patterns of surgical care and complications in elderly adults. J Am Geriatr Soc. 2014 May;62(5):829-35. doi: 10.1111/jgs.12794. Epub 2014 Apr 14. PMID 24731176
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Background] Boone MD, Sites B, von Recklinghausen FM, Mueller A, Taenzer AH, Shaefi S. Economic Burden of Postoperative Neurocognitive Disorders Among US Medicare Patients. JAMA Netw Open. 2020 Jul 1;3(7):e208931. doi: 10.1001/jamanetworkopen.2020.8931. PMID 32735336
- [Background] Oh ES, Akeju O, Avidan MS, Cunningham C, Hayden KM, Jones RN, Khachaturian AS, Khan BA, Marcantonio ER, Needham DM, Neufeld KJ, Rose L, Spence J, Tieges Z, Vlisides P, Inouye SK; NIDUS Writing Group. A roadmap to advance delirium research: Recommendations from the NIDUS Scientific Think Tank. Alzheimers Dement. 2020 May;16(5):726-733. doi: 10.1002/alz.12076. Epub 2020 Apr 14. PMID 32291901
- [Background] Goldberg TE, Chen C, Wang Y, Jung E, Swanson A, Ing C, Garcia PS, Whittington RA, Moitra V. Association of Delirium With Long-term Cognitive Decline: A Meta-analysis. JAMA Neurol. 2020 Nov 1;77(11):1373-1381. doi: 10.1001/jamaneurol.2020.2273. PMID 32658246
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126
- [Background] Fritz BA, Maybrier HR, Avidan MS. Intraoperative electroencephalogram suppression at lower volatile anaesthetic concentrations predicts postoperative delirium occurring in the intensive care unit. Br J Anaesth. 2018 Jul;121(1):241-248. doi: 10.1016/j.bja.2017.10.024. Epub 2018 Jan 17. PMID 29935578
- [Background] Pedemonte JC, Plummer GS, Chamadia S, Locascio JJ, Hahm E, Ethridge B, Gitlin J, Ibala R, Mekonnen J, Colon KM, Westover MB, D'Alessandro DA, Tolis G, Houle T, Shelton KT, Qu J, Akeju O. Electroencephalogram Burst-suppression during Cardiopulmonary Bypass in Elderly Patients Mediates Postoperative Delirium. Anesthesiology. 2020 Aug;133(2):280-292. doi: 10.1097/ALN.0000000000003328. PMID 32349072
- [Background] Soehle M, Dittmann A, Ellerkmann RK, Baumgarten G, Putensen C, Guenther U. Intraoperative burst suppression is associated with postoperative delirium following cardiac surgery: a prospective, observational study. BMC Anesthesiol. 2015 Apr 28;15:61. doi: 10.1186/s12871-015-0051-7. PMID 25928189
- [Background] Brown CH 4th, Max L, LaFlam A, Kirk L, Gross A, Arora R, Neufeld K, Hogue CW, Walston J, Pustavoitau A. The Association Between Preoperative Frailty and Postoperative Delirium After Cardiac Surgery. Anesth Analg. 2016 Aug;123(2):430-5. doi: 10.1213/ANE.0000000000001271. PMID 27096563
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Plummer GS, Ibala R, Hahm E, An J, Gitlin J, Deng H, Shelton KT, Solt K, Qu JZ, Akeju O. Electroencephalogram dynamics during general anesthesia predict the later incidence and duration of burst-suppression during cardiopulmonary bypass. Clin Neurophysiol. 2019 Jan;130(1):55-60. doi: 10.1016/j.clinph.2018.11.003. Epub 2018 Nov 16. PMID 30476711
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Besch G, Liu N, Samain E, Pericard C, Boichut N, Mercier M, Chazot T, Pili-Floury S. Occurrence of and risk factors for electroencephalogram burst suppression during propofol-remifentanil anaesthesia. Br J Anaesth. 2011 Nov;107(5):749-56. doi: 10.1093/bja/aer235. Epub 2011 Aug 8. PMID 21828343
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04713644/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04713644/ICF_000.pdf